CLINICAL TRIAL: NCT05119608
Title: Detection and Treatment of Long-term Symptoms - Post-covid Syndrome - in Patients Who Have Been Treated in Intensive Care for COVID-19.
Brief Title: Treatment of Post-covid Syndrome in Patients Treated in Intensive Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Collaborators: Region Stockholm (Other Government); Lund University (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders C Håkansson, MD, professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05128
Record Dates: First submitted 2021-11-11; First posted 2021-11-15 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Mental Health Disorder
Keywords: COVID-19; mental health disorder; cognitive-behavioral therapy; acceptance and commitment therapy; addictive behavior; ICU
MeSH Terms: conditions — COVID-19; Mental Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled trial
Masking Description: Study of a psycho-therapeutic intervention vs treatment as usual, therefore no masking of the treatment given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT/ACT (Experimental): Cognitive-behavioral therapy intervention with principal components of acceptance and commitment therapy (ACT)
  Interventions: Behavioral: CBT/ACT
- TAU (Active Comparator): Treatment as usual, defined by standard care, i.e. referral to relevant health care provider (typically primary care).
  Interventions: Behavioral: CBT/ACT

INTERVENTIONS:
Behavioral: CBT/ACT — 10-session ACT-re-enforced CBT intervention.

SUMMARY:
The present study is a pilot randomized controlled trial, which identifies and diagnoses mental health problems in survivors of critical COVID-19 infection at 12 months post-ICU care, and randomize patients to either an ACT-enforced CBT intervention, or to treatment as usual.

DETAILED DESCRIPTION:
This is a pilot RCT aiming to intervene in symptoms of poor mental health in COVID survivors at 12 months after ICU care for the COVID infection. Based on the uncertain number of patents who screen positive for mental health problems 12 months after ICU care, based on the novelty of the condition assessed, and the uncertainty about which treatment effects to expect on mental health outcomes, the study was designed as a pilot study, with feasibility measures (consent, adherence and satisfaction with the treatment) as the primary variables, and with effects on mental health symptoms as secondary variables.

The study plans to assess and randomize a convenience sample of patients, as it can not be estimated which numbers can be expected, but it is aimed to include at least 40 patients in the study (20 in the intervention group and 20 in the control group).

Specifically, the present study aims to

1. investigate early predictors (during ICU-care) of post-covid syndrome occurring at 3-6 months, 12 months, and 36 months, respectively, including cognitive and mental health problems,
2. deepen the understanding of mental health symptoms in ICU-treated COVID-19 survivors, mental health-related treatment seeking, changes in addictive behaviors, and the diagnostic meaning of mental health symptoms expressed in COVID-19 survivors, and
3. conduct a clinical treatment study with the following research question: for patients with post-covid mental health symptoms after 12 months, is an intervention of Cognitive Behavioral Therapy (CBT) with Acceptance and Commitment Therapy (ACT), when compared to standard clinical care (referral to primary care), feasible and associated with improved patient adherence and patient satisfaction, and secondly, does it improve the outcome of post-covid anxiety symptoms and secondary other symptoms of poor mental health and quality of life?

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 survivors who screen positive for clinical anxiety or depression, defined as reaching a score of ≥ 8 on either the anxiety or depression sub-scales within the questionnaire HADS at the standard 12-months follow-up

Exclusion Criteria:

* Conditions in which patients are acutely suicidal, psychotic, suffering from a mental disorder requiring in-patient psychiatric treatment, opposed to receiving a psycho-therapeutic intervention, or with cognitive problems or language difficulties which are judged to be too extensive for the informed consent procedure and for a psycho-therapeutic intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility with respect to willingness for treatment study inclusion | 8 weeks post-assessment
  Proportion of patients screened who consent to and initiate the treatment study
Feasibility with respect to patient adherence | 2 weeks post-treatment
  Proportion of patients who remain in the treatment study including complete treatment settings and 2-week follow-up
Patient satisfaction with therapy intervention | 2 weeks post-treatment
  Therapy and Therapist Scale-Revised (STTS-R)

SECONDARY OUTCOMES:
Reduction of HADS anxiety score | 2 weeks, 3 and 12 months post-treatment
  Reduction of HADS anxiety score
Reduction of HADS depression score | 2 weeks, 3 and 12 months post-treatment
  Reduction of HADS depression score
Improved mental health-related quality of life | 2 weeks, 3 and 12 months post-treatment
  Improved mental health component summary score of SF-36v2
Reduced fatigue | 2 weeks, 3 and 12 months post-treatment
  Modified Fatigue Impact Scale (MFIS)
Reduced post-traumatic symptoms | 2 weeks, 3 and 12 months post-treatment
  Posttraumatic Stress Disorder Checklist (PCL-5) scale

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Psychiatry Skåne, Malmö-Trelleborg deparment of psychiatry, Malmo
  - Södersjukhuset AB, Region Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: No